CLINICAL TRIAL: NCT01890551
Title: Dynamic Kine-mri in Patellofemoral Instability in Adolescents- an Aid in the Diagnosis
Brief Title: Kine-Mri in Patellofemoral Instability
Acronym: Knee- MRI 2012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Matti Eskelinen, professor, Kuopio University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KUH5203078
Record Dates: First submitted 2013-06-18; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Affected and Unaffected Knee in Adoloescent
Keywords: Adoloescent, patellofemoral, instability,biomechanics, magnetic resonance imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- affected knee (Other): Interest was to evaluate the patellofemoral joint biomechanics with KINE-MRI in adolescents with affected and unaffected knees in a case-control study
  Interventions: Other: Dynamic kine-mri
- unaffected knee (Other): Interest was to evaluate the patellofemoral joint biomechanics with KINE-MRI in adolescents with affected and unaffected knees in a case-control study
  Interventions: Other: Dynamic kine-mri

INTERVENTIONS:
Other: Dynamic kine-mri — Dynamic kinematic (KINE) magnetic resonance imaging (MRI) of the patellofemoral joint.

SUMMARY:
Purpose: The impact of kinematic-MRI (KINE-MRI) in the patellofemoral instability and anterior knee pain of the adolescents is rarely reported.Interest was to evaluate the patellofemoral joint biomechanics with KINE-MRI in adolescents with affected and unaffected knees in a case-control study.Methods: KINE-MRI was performed in 29 adolescents (affected knee group, AKG, n=29 and n=26 unaffected knee group, UAKG, n=26) aged 11-16 years with unilateral patellofemoral instability. For the control group invvestigators enrolled ten healthy age- and sex-matched volunteers (healthy knee group, HKG, n=19 ).The study parameters, Bisect Offset (BSO), Lateral Patellar Displacement (LPD), Patellar Tilt Angle (PTA), Sulcus Angle and Insall-Salvati ratio at 0, 10, 20 and 30 degrees of flexion-extension, were measured for the AKG patients (n=29), and UAKG patients (n=26) and the HKG subjects (n=19). Results: In a comparison between the AKG patients and the HKG subjects there was a significant difference in the BSO-ratio, LPD-test and PTA-test. In these parameters the difference between the AKG patients and the HKG subjects progressively increased towards the full extension of the knee. In the AKG and UAKG patients BSO-ratio at 0 degree ranged between 0.5 and 1.2 in both groups, whereas the BSO-ratio in the HKG subjects ranged between 0.33 and 0.75 (P < .001). At the zero degree the LPD-test ranged between 0 and 10 mm in the AKG patients and between 0 and 35 mm in the UAKG patients, whereas the lateral displacement-test ranged between 0 and 5 mm in the HKG subjects (P = .003). Patellar tilt angle-test ranged between -30 and 20 degrees in the AKG patients and between -30 and 24 degrees in the UAKG patients and in the HKG subjects the PTA-test ranged between 10 and 24 degrees (P < .001).Conclusion: The KINE-MRI could be a feasible method for the evaluation of patellar tracking in adolescents.

DETAILED DESCRIPTION:
Purpose: The impact of kinematic-MRI (KINE-MRI) in the patellofemoral instability and anterior knee pain of the adolescents is rarely reported.Interest was to evaluate the patellofemoral joint biomechanics with KINE-MRI in adolescents with affected and unaffected knees in a case-control study.Methods: KINE-MRI was performed in 29 adolescents (affected knee group, AKG, n=29 and n=26 unaffected knee group, UAKG, n=26) aged 11-16 years with unilateral patellofemoral instability. For the control group investigators enrolled ten healthy age- and sex-matched volunteers (healthy knee group, HKG, n=19 ).The study parameters, Bisect Offset (BSO), Lateral Patellar Displacement (LPD), Patellar Tilt Angle (PTA), Sulcus Angle and Insall-Salvati ratio at 0, 10, 20 and 30 degrees of flexion-extension, were measured for the AKG patients (n=29), and UAKG patients (n=26) and the HKG subjects (n=19). Results: In a comparison between the AKG patients and the HKG subjects there was a significant difference in the BSO-ratio, LPD-test and PTA-test. In these parameters the difference between the AKG patients and the HKG subjects progressively increased towards the full extension of the knee. In the AKG and UAKG patients BSO-ratio at 0 degree ranged between 0.5 and 1.2 in both groups, whereas the BSO-ratio in the HKG subjects ranged between 0.33 and 0.75 (P < .001). At the zero degree the LPD-test ranged between 0 and 10 mm in the AKG patients and between 0 and 35 mm in the UAKG patients, whereas the lateral displacement-test ranged between 0 and 5 mm in the HKG subjects (P = .003). Patellar tilt angle-test ranged between -30 and 20 degrees in the AKG patients and between -30 and 24 degrees in the UAKG patients and in the HKG subjects the PTA-test ranged between 10 and 24 degrees (P < .001).Conclusion: The KINE-MRI could be a feasible method for the evaluation of patellar tracking in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the 29 patients were as follows: objective patellar instability with or without objective or episodic patellar dislocation, anterior knee pain for more than one year with positive apprehension tests, J-tracking of the patella, lateral tilt and displacement proven clinically.

Exclusion Criteria:

* did not enroll any patients with the knee trauma, the previous surgery and the osteochondritic lesions.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 1998-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Bisect Offset (BSO) | One year
  BSO is the ratio of medial to lateral displacement of the patella (Brossmann et al. Radiology 1993).

SECONDARY OUTCOMES:
Lateral Patellar Displacement (LPD) | One year
  LPD is the lateral displacement of the patella.
Patellar Tilt Angle (PTA) | One year
  PTA measures the lateral tilting of the patella.
Sulcus Angle | One year
  Sulcus Angle measures the angle formed by the medial and lateral borders of the trochlea
Insall-Salvati-ratio | One year
  Insall-Salvati-ratio measures the ratio of the length of the patella to the length of the patellar ligament.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Eskelinen, professor, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland